CLINICAL TRIAL: NCT00252447
Title: A Pilot Study of Pre-Operative Conformal Radiotherapy in Patients With Radical Prostatectomy
Brief Title: Preop Conformal Radiotherapy - Prostate
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 01-0483-C
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Last update posted 2010-08-11 (Estimated); Status verified 2010-08

CONDITIONS: Prostatic Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms

INTERVENTIONS:
Procedure: Pre-Operative Conformal Radiotherapy

SUMMARY:
Radical prostatectomy and radical radiation therapy remain the standard treatment approaches for patients with clinically localized prostate cancer (T1, T2).Radical prostatectomy is most effective when the disease is organ confined at the time of surgery. However, in many series up to 60% of patients have positive resection margins at the time of surgery and there is evidence to suggest that these patients may not be curable by surgery alone. A number of preoperative clinical variables including clinical stage, serum Prostate Specific Antigen (PSA) and Gleason scorea re helpful in determining the probability of finding organ confined disease at the time of syrgery.

ELIGIBILITY:
* Histologically confirmed carcinoma of the prostate
* High risk localized disease defined as clinical T1 or T2 plus [ (i) Gleason ¡Ý7, PSA>10 ng/ml and <35 ng/ml OR (ii) PSA >15 ng/ml and less <35 ng/ml (any Gleason) ]
* No evidence of pelvic lymph node metastases on CT scan within 4 months of surgery
* No evidence of distant metastases on bone scan within 4 months of surgery
* No contraindication to pelvic radiation therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15
Dates: Start 2000-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To document the feasibility of pre-operative conformal radiation therapy in patients undergoing radical prostatectomy for localized prostate cancer who are at high risk for having local extra-prostatic disease at time of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Padraig Warde, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- University Health Network Princess Margaret Hospital, Toronto, Ontario, Canada